CLINICAL TRIAL: NCT02260635
Title: A Double-Blind Efficacy and Safety Study of Evacetrapib Followed by an Open-Label Extension in Japanese Patients With Primary Hypercholesterolemia
Brief Title: A Study of Evacetrapib (LY2484595) in Japanese Participants With Primary Hypercholesterolemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study termination due to insufficient efficacy.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14503; I1V-JE-EIBI (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — evacetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evacetrapib (Experimental): 130 milligrams (mg) evacetrapib given orally (PO) once a day for 12 weeks. Participants begin open label extension (130 mg evacetrapib given orally once a day for 40 weeks) after week 12.
  Interventions: Drug: Evacetrapib
- Placebo (Placebo Comparator): Placebo given PO once a day for 12 weeks. Participants begin open label extension (130 mg evacetrapib given PO once a day for 40 weeks) after week 12.
  Interventions: Drug: Evacetrapib; Drug: Placebo

INTERVENTIONS:
Drug: Evacetrapib — Administered orally
  Other Names: LY2484595
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of the study drug known as evacetrapib in Japanese participants with primary hypercholesterolemia. The double blind treatment period will last for 12 weeks and the open-label extension period will last for an additional 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Japanese outpatients who are diagnosed with primary hypercholesterolemia with LDL-C levels (measured by a direct method at baseline) that meet the following criteria. (Participant categories are based on the definition in Japan Atherosclerosis Society 2012 guidelines.)

  * Category I: 160 mg/deciliter (dL)≤LDL-C<200 mg/dL
  * Category II: 140 mg/dL≤LDL-C<175 mg/dL
  * Category III: 120 mg/dL≤LDL-C<150 mg/dL
* Have triglycerides (TG) ≤400 mg/dL.
* Have HDL-C <100 mg/dL.

Exclusion Criteria:

* Participants on LDL apheresis or plasma apheresis.
* Participants with secondary hypercholesterolemia or familial hypercholesterolemia.
* Any planned angiography. If angiography is planned, participants may be screened and enrolled after all such planned procedures are completed.
* History of any of the following any conditions:

  * Stable angina or acute coronary syndrome (unstable angina, myocardial infarction), old myocardial infarction or a coronary revascularization procedure including stent placement, or symptomatic carotid artery disease
  * peripheral arterial disease
  * ischemic stroke or transient ischemic attack (TIA)
  * intracranial hemorrhage
  * abdominal aortic aneurysm
* Have systolic blood pressure (SBP) >160 millimeters of mercury (mm Hg) or diastolic blood pressure (DBP) >100 mm Hg.
* Have a hemoglobin A1c ≥8.4% (National Glycohemoglobin Standardization Program).
* During the study period, participants who plan to use, are likely to require, or unwilling or unable to stop with adequate washout any prescription, over the counter medication, supplements or health foods with the intent to treat serum lipids (LDL-C, HDL-C, TG) including but not limited to these classes of drugs: statin, ezetimibe, bile acid sequestrant, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). Participants taking probucol, fibrate or nicotinic agents within 8 weeks before screening are excluded from the study.
* Have been exposed to cholesteryl ester transfer protein inhibitors (e.g., anacetrapib or dalcetrapib).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo given PO once a day for 12 weeks. Participants begin open label extension (130 mg evacetrapib given orally once a day for 40 weeks) after week 12.
Period: Double-Blind Treatment Period
Arm/Group | Evacetrapib | Placebo
Started | 27 | 27
Received at Least One Dose of Study Drug | 27 | 26
Completed | 26 | 25
Not Completed | 1 | 2
Not completed — Failure to Meet Randomization Criteria | 1 | 2
Period: Open-Label Extension
Arm/Group | Evacetrapib | Placebo
Started | 26 | 25
Received at Least One Dose of Study Drug | 26 | 25
Completed | 0 | 0
Not Completed | 26 | 25
Not completed — Study Termination | 25 | 25
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Evacetrapib: 130 milligrams (mg) evacetrapib given orally once a day for 12 weeks. Participants begin open label extension (130 mg evacetrapib given orally once a day for 40 weeks) after week 12.
- Placebo: Placebo given orally once a day for 12 weeks. Participants begin open label extension (130 mg evacetrapib given orally once a day for 40 weeks) after week 12.
- Total: Total of all reporting groups
Arm/Group | Evacetrapib | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (10.19) | 53.3 (10.13) | 52.8 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 20 | 17 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 27 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 in Low-Density Lipoprotein Cholesterol (LDL-C) Measured by Beta Quantification
Description: Least Square Mean (LS mean) using mixed model repeated measures (MMRM) adjusted for baseline, treatment, visit , and treatment*visit, where the participant is a random effect.
Time Frame: Baseline, Week 12
Population: All randomized participants receiving at least 1 dose of study drug with evaluable LDL-C values measured by beta quantification at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percent change in LDL-C
Groups:
- Evacetrapib: 130 milligrams (mg) evacetrapib given PO once a day for 12 weeks. Participants begin open label extension (130 mg evacetrapib given PO once a day for 40 weeks) after week 12.
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 26 | 25
percent change in LDL-C | -34.27 (3.908) | 0.00 (3.984)

2. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C)
Description: LS mean using MMRM adjusted for baseline, treatment, visit , and treatment*visit, where the participant is a random effect.
Time Frame: Baseline, Week 12
Population: All randomized participants receiving at least 1 dose of study drug with evaluable HDL-C values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percent change of HDL-C
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 26 | 25
percent change of HDL-C | 123.57 (6.697) | -0.45 (6.805)

3. Secondary Outcome: Percent Change From Baseline in LDL-C (Direct)
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: All randomized participants receiving at least 1 dose of study drug with evaluable LDL-C direct values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percent change of LDL-C direct
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 26 | 25
percent change of LDL-C direct | -33.86 (3.163) | 0.22 (3.226)

4. Secondary Outcome: Percent Change From Baseline in Non HDL-C
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: All randomized participants receiving at least 1 dose of study drug with evaluable Non HDL-C values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percent change in non HDL-C
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 26 | 25
percent change in non HDL-C | -26.48 (3.171) | -0.03 (3.237)

5. Secondary Outcome: Percent Change From Baseline in Lipoprotein-a
Description: LS Mean from analysis of covariance (ANCOVA) model adjusted for baseline and treatment.
Time Frame: Baseline, Week 12, Week 52
Population: All randomized participants receiving at least 1 dose of study drug with evaluable Lipoprotein-a values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percent change in Lipoprotein-a
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 17 | 24
percent change in Lipoprotein-a
  Week 12 | -35.71 (6.574) | 3.54 (5.532)
  Week 52 | NA (NA) — Week 52 data not available due to early termination of this study. | NA (NA) — Week 52 data not available due to early termination of this study.

6. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-I
Description: LS Mean from ANCOVA model adjusted for baseline and treatment.
Time Frame: Baseline, Week 12, Week 52
Population: All randomized participants receiving at least 1 dose of study drug with evaluable Apolipoprotein A-I values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percent change in Apolipoprotein A-I
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 27 | 26
percent change in Apolipoprotein A-I
  Week 12 | 49.1 (3.44) | -2.5 (3.51)
  Week 52 | NA (NA) — Week 52 data not available due to early termination of this study. | NA (NA) — Week 52 data not available due to early termination of this study.

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B
Description: LS Mean from ANCOVA model adjusted for baseline and treatment.
Time Frame: Baseline, Week 12, Week 52
Population: All randomized participants receiving at least 1 dose of study drug with evaluable Apolipoprotein B values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percent change in Apolipoprotein B
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 27 | 26
percent change in Apolipoprotein B
  Week 12 | -29.0 (2.65) | -1.3 (2.70)
  Week 52 | NA (NA) — Week 52 data not available due to early termination of this study. | NA (NA) — Week 52 data not available due to early termination of this study.

ADVERSE EVENTS:
Description: All randomized participants who received at least 1 dose of study drug.
Groups:
- Evacetrapib Double Blind Treatment Period: 130mg evacetrapib given PO once a day for 12 weeks.
- Placebo Double Blind Treatment Period: Placebo given PO once a day for 12 weeks
- Evacetrapib Open Label Extension; Placebo/Evacetrapib Open Label Extension: Participants begin open label extension (130 mg evacetrapib given PO once a day for 40 weeks) after week 12.
Arm/Group | Evacetrapib Double Blind Treatment Period | Placebo Double Blind Treatment Period | Evacetrapib Open Label Extension | Placebo/Evacetrapib Open Label Extension
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 5/27 | 7/26 | 6/26 | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evacetrapib Double Blind Treatment Period (N=27) | Placebo Double Blind Treatment Period (N=26) | Evacetrapib Open Label Extension (N=26) | Placebo/Evacetrapib Open Label Extension (N=25)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 3 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza b virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to anticipated Inefficient efficacy of the I1V-MC-EIAN (NCT01687998) study, therefore Week 52 data is not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days